CLINICAL TRIAL: NCT01739504
Title: An Open-label, Non-Randomized, Multi-Center Study to Assess the Safety and Effects of Autologous Adipose-Derived Stromal Cells Delivered Intra- Articularly in Patients With Osteoarthritis
Brief Title: Autologous Adipose-Derived Stromal Cells Delivered Intra-articularly in Patients With Osteoarthritis.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: company dissolved
Sponsor: Ageless Regenerative Institute (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AD-US-OR-001
Record Dates: First submitted 2012-09-28; First posted 2012-12-03 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2016-09

CONDITIONS: Osteoarthritis
Keywords: Arthritis; Joint pain; Articular cartilage; Mesenchymal stem cells; Autologous; Adipose tissue
MeSH Terms: conditions — Osteoarthritis; Arthritis; Arthralgia | interventions — Lipectomy; Anesthesia, Local

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autologous Adipose-derived Stromal Vascular Fraction infusion (Experimental): Intervention: AD-SVF infusion directly into affected joints.
  Interventions: Procedure: Liposuction with Local Anesthesia; Biological: Intra articular infusion of AD-SVF

INTERVENTIONS:
Procedure: Liposuction with Local Anesthesia — Liposuction under tumescent anesthesia for adipose tissue harvesting.
  Other Names: Lipoplasty; Liposculpture; Suction-assisted fat removal
Biological: Intra articular infusion of AD-SVF — Adipose tissue is available in most patients for harvest through minimally invasive procedures such as liposuction. AD-SVF can be obtained in large quantities after processing of adipose tissue in the laboratory.
  * AD-SVF to promote tissue regeneration and repair with their ability to secrete various growth factors that can modulate host tissue environment.
  * Patient's AD-SVF combined with PRP are used for direct intra-articular injection after processing.

SUMMARY:
This will be an open-label, non-randomized, multi-center, patient sponsored study of Adipose-Derived Stromal Vascular Fraction (AD-SVF) implantation performed intra-articularly to affected joints.

The intent of this clinical study is to answer the questions: 1) Is the proposed treatment safe and 2) Is treatment effective in improving the disease pathology of patients with diagnosed Osteoarthritis.

DETAILED DESCRIPTION:
AD-SVF will be collected from the patient's adipose-derived tissue (body fat). Using local anesthesia, Liposuction will be performed to collect the adipose tissue specimen. The adipose tissue is then transferred to the laboratory for separation of AD-SVF. In addition, patient's peripheral blood will be collected for isolation of platelet rich plasma (PRP), which are then combined with the AD-SVF for intra-articular administration of affected joint.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females between Age 18 and 80 years.
* Patient with current proven diagnosis of Osteoarthritis, with consistent symptomatology
* Up to date on all age and gender appropriate cancer screening per American Cancer Society.

Exclusion Criteria:

* Females who are pregnant or nursing or females of childbearing potential who are unwilling to maintain contraceptive therapy for the duration of the study.
* Life expectancy < 6 months due to concomitant illnesses.
* Exposure to any investigational drug or procedure within 1 month prior to study entry or enrolled in a concurrent study that may confound results of this study.
* Active infectious disease. Patients known to have tested positive for HIV, HTLV, HBV, HCV, CMV (IgM > IgG) and/or syphilis will have an expert consultation as to patient eligibility based on the patient's infectious status
* Any illness which, in the Investigator's judgment, will interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of the study results
* Patients on chronic immunosuppressive transplant therapy
* Systolic blood pressure (supine) ≤90 mm Hg or greater than 180mmHg
* Resting heart rate > 100 bpm;
* Known drug or alcohol dependence or any other factors which will interfere with the study conduct or interpretation of the results or who in the opinion of the investigator are not suitable to participate.
* History of cancer (other than non-melanoma skin cancer or in-situ cervical cancer) in the last five years.
* Active clinical infection
* Unwilling and/or not able to give written informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Visual Analogue Scale (VAS) | 3 months, 6 months
  For pain score, functional rating index, visual analog scale (VAS), physical therapy (PT), and range of motion (ROM) were determined as previously described. The patient was restricted from taking steroids, aspirin, nonsteroidal anti-inflammatory drugs (NSAIDs) for one week prior to the procedure.
Change from Baseline of Quality of life scores | 3 months, and 6 months
Change from Baseline of Reduction in analgesics | Baseline, 3 months, 6 months
Number of adverse events reported | 6 months

SECONDARY OUTCOMES:
Change from Baseline in x-ray, sonogram, or MRI imaging of affected joint compared to baseline. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sharon McQuillan, MD, Principal Investigator — Ageless Regenerative Institute
Locations (1):
- Ageless Institute LLC, Aventura, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided